CLINICAL TRIAL: NCT04578197
Title: NeuroCOVID - A Study of Activation and Inhibition of the Immune and Coagulation Systems, the Presence of Biochemical (Blood / CSF) and Structural Brain Changes and Their Association With Long-term Cognitive Dysfunction in Intensive Care-requiring Covid-19 Patients
Brief Title: NeuroCovid - a Study of Intensive Care-requiring Covid-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Lars I Eriksson, Professor, Karolinska University Hospital
Other Study IDs: Dnr 2020-02760
Record Dates: First submitted 2020-09-02; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: SARS-CoV-2; intensive care; neurocognitive disorders; cognitive dysfunction; biochemical and structural brain changes
MeSH Terms: conditions — COVID-19; Neurocognitive Disorders; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Critically ill patients requiring intensive care suffer to a large extent from cognitive deficits involving higher brain functions that primarily affect memory, learning and the ability to concentrate. While the background to this effect is not fully understood, there are growing evidence to support mechanisms related to neuro inflammation and changes in blood flow with concomitant ischemic brain damage. Patients with covid-19 often suffer from severe inflammatory activity with an increased risk of coagulation abnormalities and brain damage. Covid-19 patients requiring intensive care develope more severe impairment of neurological and cognitive function than critically ill intensive care patients who have not covid-19. This project therefore aims to map the link between inflammation, immunology and coagulation systems as well as biochemical and structural changes in the brain with cognitive effects in patients in intensive care for covid-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Need for Intensive care
* Positive PCR test for SARS-CoV-2

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 50 women and 50 men
Study Population: Men and women with covid-19 (positive PCR test for Coronavirus SARS-CoV-2 RNA) who are admitted to the Intensive Care Unit at Karolinska University Hospital in Solna and Huddinge
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-18 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
The association between changes in blood biomarkers for inflammation and the presence of neuroradiologically verified brain injury and neurocognitive disorder | Up to 12 months
The association between changes in blood biomarkers for nerve cell damage and the presence of neuroradiologically verified brain injury and neurocognitive disorder | Up to 12 months
The association between changes in blood biomarkers for neurodegeneration and the presence of neuroradiologically verified brain injury and neurocognitive disorder | Up to 12 months

SECONDARY OUTCOMES:
The association between changes in coagulation factors and the presence of neuroradiologically verified brain injury and / or neurocognitive disorder | Up to 12 months
The association between changes in coagulation ability (ROTEM analysis - rotational thromboelastometry) and the presence of neuroradiologically verified brain injury and / or neurocognitive disorder | Up to 12 months
The association between changes in inflammatory biomarkers and the presence of neuroradiologically verified brain injury and / or neurocognitive disorder | Up to 12 month
Blood biomarker changes of inflammation impact | Up to 3 months
  Markers of inflammation impact - in relation to cerebrospinal fluid changes .
Blood biomarker changes of neurological impact | Up to 3 months
  Markers of neurological impact - in relation to cerebrospinal fluid changes .
Neuroradiological changes | Up to 3 months
  Neurological impact in relation to cerebrospinal fluid changes
Clinical course - Pulmonary gas exchange | Up to 3 months
  in relation to cerebrospinal fluid changes/blood
Clinical course - Lung function recording | Up to 3 months
  in relation to cerebrospinal fluid changes/blood
Patient characteristics | Up to 3 months
  Patient ICU care data - in relation to cerebrospinal fluid changes

CONTACTS AND LOCATIONS:
Overall Officials: Lars I Eriksson, Professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden